CLINICAL TRIAL: NCT02796313
Title: Diet Intervention for Hypertension: Adaptation and Dissemination to Native Communities
Acronym: NOSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: Oklahoma State University (Other)
Responsible Party: Principal Investigator, Dedra Buchwald, Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01HL126578 (NIH)
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will receive tailored advice on adopting a low-sodium DASH diet, comprising nutritional education and ongoing guidance for purchasing heart-healthy foods, plus a weekly $35 credit for groceries.
  Interventions: Behavioral: DASH Groceries + Weekly Sessions
- Control Group (Active Comparator): Participants in the control group will receive printed educational materials with general information about low-salt diets plus a weekly $35 credit for groceries.
  Interventions: Behavioral: Groceries + Brochure

INTERVENTIONS:
Behavioral: DASH Groceries + Weekly Sessions — Intervention group participants will receive 1 hour of in-person nutritional counseling and a personalized prescription for the low-salt DASH diet based on estimated calorie needs at baseline, followed by weekly 20-minute phone calls in weeks 1-8 to provide extra support.
  Arms: Intervention Group
Behavioral: Groceries + Brochure — Control group participants will receive a printed brochure about the health benefits of a low-salt diet. They will place an unrestricted $35 grocery order for 8 weeks.
  Arms: Control Group

SUMMARY:
We will conduct a randomized trial to test our DASH (Dietary Approaches to Stop Hypertension) based intervention in 370 adult American Indians with inadequately controlled systolic blood pressure (≥130 mmHg). Over the 5 years of the project, we will recruit and randomize 200 participants from each of 4 urban sites: two in Washington, one in Oklahoma, and one in South Dakota.

DETAILED DESCRIPTION:
All participants complete 3 data collection visits following an over-the-phone eligibility screening call (baseline, week 8, and week 12). Participants will be randomized into either the control group or the intervention group at the baseline visit.

All participants will receive 8 weekly credits for groceries and will be given equipment for monitoring their BP at home. Study staff will help participants place their grocery orders each week, and will collect readings from the home BP monitoring equipment at the same time. This data will be used to understand whether the intervention is effective for controlling BP.

All participants will be encouraged to maintain their regular levels of physical activity and receive treatment as usual from their healthcare providers.

The control group participants will receive an American Heart Association printed brochure about the health benefits of a low-salt diet. All foods will be available to purchase, including those that do not meet the DASH diet guidelines.

The intervention group participants will receive 1 hour of nutritional counseling over the phone and a personalized prescription for the low-salt DASH diet based on estimated calorie needs at baseline, followed by weekly 20-minute phone calls in weeks 1-8 to provide extra support.

The intervention group's food choices will be limited to fresh produce and a pre-determined list of other foods included in the DASH diet. During weekly phone calls, the dietitian will use a structured phone curriculum to discuss in more detail a different component of the DASH diet, followed by goal setting related to that component. Through small goal setting each week, participants will receive ongoing support to improve full adherence to the DASH diet by the end of week 8.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* be at least 18 years old;
* have had diagnosed hypertension for at least 1 year;
* be on a stable routine of antihypertensive medications for at least 2 months OR not currently medicated, without anticipated changes for the duration of the study;
* have systolic BP ≥ 130 mmHg at the past 2 clinic visits and at the screening call;
* have access to regular medical care and permission from their primary care provider to participate (study staff obtain verbal permission before recruiting participants);
* be physically and cognitively able to use the home BP monitoring device;
* be willing and able to follow all other study procedures.

Exclusion Criteria:

People are ineligible if they:

* experienced incident cardiovascular disease or stroke within the previous 6 months;
* have a known diagnosis of secondary hypertension (e.g., renal artery stenosis);
* have a recent history of high blood potassium due to certain medications that can raise potassium levels;
* have diagnosed Stage 4 or 5 kidney disease;
* are currently or planning to become pregnant during the course of the study;
* are participating in another health research study involving hypertension;
* are receiving treatment for cancer or another serious or terminal medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-04 (Actual)

PRIMARY OUTCOMES:
Improved blood pressure | 12 weeks
  Systolic blood pressure measurements collected throughout the study.

SECONDARY OUTCOMES:
Improved urinary sodium/potassium levels | 12 weeks
  Measured by 24 hour urine samples collected at 3 time points.
Improved BMI | 12 weeks
  Measured by weight and height. Waist circumference will also be measured.
Improved blood lipids | 12 weeks
  Measured by cholesterol panel at 3 time points

CONTACTS AND LOCATIONS:
Overall Officials: Dedra Buchwald, Principal Investigator — Washington State University
Locations (4):
- United States (4):
  - Chickasaw Nation Health Clinic, Purcell, Oklahoma
  - Avera Research Institute, Rapid City, South Dakota
  - Seattle Indian Health Board, Seattle, Washington
  - NATIVE Project, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sinclair K, Nguyen CJ, Wetherill MS, Nelson K, Jackson AM, Taniguchi T, Jernigan VBB, Buchwald D. Native opportunities to stop hypertension: study protocol for a randomized controlled trial among urban American Indian and Alaska Native adults with hypertension. Front Public Health. 2023 Jun 2;11:1117824. doi: 10.3389/fpubh.2023.1117824. eCollection 2023. PMID 37333529